CLINICAL TRIAL: NCT00939133
Title: Double Blinded Vehicle Controlled Proof of Concept Study to Investigate the Recurrence of Inflammatory and Non-inflammatory Acne Lesions Using Tretinoin Gel (Microsphere) 0.04% in Male Patients Post Oral Isotretinoin Use
Brief Title: Proof of Concept Study to Investigate the Recurrence of Acne Post Isotretinoin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dermatrials Research (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Ronald Vender MD FRCPC, MD FRCPC, Dermatrials Research
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: C2009-01
Record Dates: First submitted 2009-07-11; First posted 2009-07-14 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Acne
Keywords: acne; tretinoin; isotretinoin; recurrence; Retin A micro
MeSH Terms: conditions — Acne Vulgaris; Recurrence | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tretinoin microsphere 0.04% gel (Active Comparator)
  Interventions: Drug: tretinoin microsphere 0.04% gel
- Vehicle gel (Placebo Comparator)
  Interventions: Drug: vehicle gel

INTERVENTIONS:
Drug: tretinoin microsphere 0.04% gel — Applied daily to entire face for six months
  Other Names: Retin A micro 0.04%
  Arms: Tretinoin microsphere 0.04% gel
Drug: vehicle gel — Placebo
  Arms: Vehicle gel

SUMMARY:
The use of topical retinoids is a mainstay and basis of early acne treatment to prevent the progression to inflammatory lesions. Post oral isotretinoin, it is not uncommon for non-inflammatory papules and comedones to recur. However, there has been no formal study to look at the prevention of recurrence of these acne lesions post isotretinoin in a long term basis. This may enhance the therapeutic options for post isotretinoin patients in order to prevent recurrence of their disease.

Hypothesis Tretinoin microsphere 0.04% will prevent recurrence of acne lesions.

DETAILED DESCRIPTION:
Subjects will be randomized 1:1 to study product or vehicle. Subjects will be randomly assigned to each group by an unblinded dispenser.

The study duration will be 24 weeks with visits at baseline (week 0), week 4, week 8, week 16 and week 24. All study products will be administered once daily for 24 weeks. Subjects will apply a sufficient amount of study product to cover the entire face.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria to be eligible for study admission:

* Males aged between 18 and 45 years old who have successfully completed a treatment of acne with oral isotretinoin (Min 4 months/Maximum 6 months with an average of 5 months and a total of 120-150mg/kg/course).
* Who can attend scheduled study follow-up visits at the outpatient dermatology clinic.
* Agree to informed consent for participation in a study.
* Agree to comply with the treatment and follow up procedures.

Exclusion Criteria:

* Patients who receive isotretinoin for condition other than acne vulgaris.
* Patients who have been off isotretinoin for less than 30 days or more than 90 days at the time of enrollment of the study.
* Patients who have used prescription topical acne treatment (tretinoin, benzoyl peroxide, topical antibiotics or any combination products) between the end of therapy of isotretinoin within 2 weeks of study enrollment or oral antibiotics of any type between the end of therapy of isotretinoin within 4 weeks of study enrollment and throughout the study.
* Patients who have been previously diagnosed with an endocrinological disorder likely to cause acne such as genital/adrenal hyperplasia, adrenal tumors or any other hypo androgenetic state.
* Patients who are using any of the systemic medications likely to cause or abate acne such as oral Dilantin or any other epileptic, Finasteride, Spironolactone or Flutamine, testosterone or dietary body-building protein powders.
* Have any nodulo-cystic lesions at baseline.
* Used topical corticosteroids on the face or systemic corticosteroids within the past 4 weeks. Use of inhaled, intra-articular, or intra-lesional steroids other than for facial acne is acceptable.
* Are currently using any medication that in the opinion of the investigator may affect the action or evaluation of the study product or place the subject at undue risk.
* Used abradants, facials, peels containing glycolic or other acids; masks, washes, or soaps containing BPO, salicylic acid, or sulfacetamide sodium; non-mild facial cleansers; moisturizers that contain retinol, salicylic acid, or α- or β-hydroxy acids within the past 2 weeks.
* Plan to use medications that are reported to exacerbate acne (e.g., mega-doses of certain vitamins, such as vitamin D [> 2000 IU per day] and vitamin B12 [> 1 mg/day], haloperidol, halogens [e.g., iodide and bromide], lithium, hydantoin, and phenobarbital), because these may impact efficacy assessments. Subjects who plan to use multivitamins, iron supplements and folate are acceptable.
* Had a facial procedure (such as chemical or laser peel, microdermabrasion, blue light treatment, etc) performed by an esthetician, beautician, physician, nurse, or other practitioner, within the past 4 weeks or if it is planned to be performed during the conduct of the study.
* Have a known hypersensitivity or have had previous allergic reaction to any of the active components or excipients of the study product.
* Used any investigational therapy within the past 4 weeks, or currently participating in another clinical study.
* Are currently abusing drugs or alcohol (drug screening not required).
* Have a significant medical history of being immunocompromised.
* Have other conditions that, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study.
* Had any major illness within 30 days before the screening examination.
* Currently are employees of R Vender, an investigator, or contract research organization (CRO) involved in the study, or an immediate family member (partner, offspring, parents, siblings or sibling's offspring) of an employee involved in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Primary objectives-to assess the efficacy of Retin A micro 0.04% on the recurrence rate of acne post isotretinoin use compared to vehicle. | Six Months

SECONDARY OUTCOMES:
The percent change in lesion counts from baseline to week 16 and 24. | Six Months
Proportion of subjects who have a Subject's Global | Assessment score of 0 or 1 at week 16 and 24
Proportion of subjects who have an ISGA score of 0 or 1 at week 16 and 24. | At week 16 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Vender, MD FRCPC, Principal Investigator — Dermatrials Research
Locations (1):
- Dermatrials Research, Hamilton, Ontario, Canada